CLINICAL TRIAL: NCT07148570
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on Pain, Comfort, and Physiological Parameters in Newborns Delivered Vaginally in the Delivery Room
Brief Title: The Effect of Nursing Care Based on Kolcaba Comfort Theory in the Delivery Room
Acronym: kolcaba Comfor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Fahri AŞKAN, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FASKAN
Record Dates: First submitted 2025-08-18; First posted 2025-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Comfort; Pain
Keywords: Kolcaba Comfort Theory; pain; Delivery room
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Participant group (Experimental): During the implementation process, neonates in the experimental group will receive care in line with Kolcaba's comfort theory throughout their stay in the intensive care unit..
  Interventions: Other: Nursing Care Based on Kolcaba's Comfort Theory
- Control group (No Intervention): In this study, the control group will receive standard care

INTERVENTIONS:
Other: Nursing Care Based on Kolcaba's Comfort Theory — Delivery Room Nursing Care Based on Kolcaba's Comfort Theory
  Arms: Experimental: Participant group

SUMMARY:
Newborns may experience pain, stress, and physiological changes during and after birth. Appropriate nursing care during this period can reduce negative effects by increasing the baby's comfort. Kolbaba's Comfort Theory aims to provide holistic care by supporting physical, psychological, environmental, and sociocultural comfort. This study aims to investigate the effects of nursing interventions based on Kolcaba's theory on pain, comfort, crying duration, and physiological parameters (heart rate, respiratory rate, SpO₂, body temperature, etc.) in noenates delivered vaginally. The findings aim to reveal the contribution of comfort-focused approaches in noenates care to clinical outcomes.

DETAILED DESCRIPTION:
Newborns may experience pain, stress, and physiological changes during and after birth. Appropriate nursing care during this period can reduce negative effects by increasing the baby's comfort. Kolbaba's Comfort Theory aims to provide holistic care by supporting physical, psychological, environmental, and sociocultural comfort. This study aims to investigate the effects of nursing interventions based on Kolcaba's theory on pain, comfort, crying duration, and physiological parameters (heart rate, respiratory rate, SpO₂, body temperature, etc.) in noenates delivered vaginally. The findings aim to reveal the contribution of comfort-focused approaches in noenates care to clinical outcomes.

Kolcaban's Comfort Theory for Care in the Delivery Room

Intervention Group:

1. Physical sub-dimension; 2. Psychospiritual comfort sub-dimension: White noise playback; skin-to-skin contact; gentle touch; 3. Sociocultural comfort sub-dimension: Family-centered care (providing contact with parents), respect for cultural practices; 4. Care will be provided in accordance with the Environmental Comfort sub-dimension..

Research Population and Sample: The study will be conducted on newborns born vaginally in the maternity ward and whose parents are eligible and agree to participate in the study. Sample: This study will be conducted on newborns selected on a voluntary basis, meeting the inclusion criteria, gestational age 38-42 weeks, 2500-4000 g, and an Apgar score ≥7. Sample Size: The number determined by power analysis, e.g., 60 infants (30 experimental, 30 control).

Study Inclusion Criteria: The baby was born vaginally; the gestational age was 38 weeks or older; the baby had no congenital anomalies; the baby had a Power (1-β err prob); the baby was breathing spontaneously; the baby did not require oxygen support; the baby was a singleton; the baby had an Apgar score between 7 and 10 at the 1st and 5th minutes; The first invasive procedure was the administration of vitamin K and hepatitis B vaccine; the same researcher performed the intramuscular injection on each baby; no assistive equipment was used during birth; and the family agreed to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery newborns in the delivery room
* Spontaneous vaginal delivery
* Stable condition (APGAR ≥7 at 5 minutes)
* No congenital anomalies
* Gestational age ≥37 weeks
* Birth weight ≥2500g
* No maternal sedation/analgesia in last 4 hours
* No neonatal resuscitation required

Exclusion Criteria:

* Preterm infants (<37 weeks)
* Maternal fever (>38°C) or chorioamnionitis
* Major congenital anomalies
* Need for NICU admission
* Maternal general anesthesia

Ages: 0 Hours to 4 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
COMFORTneo Scale | From the starting point to at least the second hour
  The COMFORTneo scale is a validated Likert-type tool assessing neonatal comfort, pain, and distress through six behavioral parameters (facial tension, muscle tone, crying, alertness, calmness/agitation, respiratory response, and body movements). Scores range from 6 (optimal comfort) to 30 (severe distress), with 4-6 indicating moderate and 7-10 severe pain/distress (van Dijk et al., 2005).
Neonatal Pain Scale | From the starting point to at least the second hour
  The NIPS uses 1 physiological (respiratory pattern) and 5 behavioral parameters (crying, alertness, facial expression, arm/leg movements) to assess pain in newborns. The scale is scored from 0 to 7, with higher scores indicating severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided